CLINICAL TRIAL: NCT02359760
Title: Assessment of Piezoelectric Periodontal Surgery Effects on Orthodontic Treatment: a Prospective Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Clarice Nishio, Ph.D, Université de Montréal
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMontreal
Record Dates: First submitted 2015-02-04; First posted 2015-02-10 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Malocclusion
Keywords: Rapid orthodontics; accelerated orthodontics; Piezocision; flapless corticotomies; minimaly invasive
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Piezocision group (Experimental): The experimental group will consist of 14 adults, subjects from 18 to 40 years-old (10 women, 4 men).
  Interventions: Procedure: Piezocision
- conventional orthodontics (No Intervention): The control group will consist of 30 matched patients with the same inclusion and exclusion criteria, who have been already treated by conventional orthodontics in the orthodontic clinic of the University of Montreal.

INTERVENTIONS:
Procedure: Piezocision — Flapless corticotomies
  Arms: Piezocision group

SUMMARY:
INTRODUCTION: Dentoalveolar surgeries such as piezocision, have been developed with the aim to accelerate the tooth movement and therefore reduce the length of orthodontic treatment. Although this surgical technique seems to present several advantages, such as decreased risk of decalcification or orthodontic relapse, its use as a routine practice is not yet recommended. The main purpose of this study is to determine the duration of orthodontic treatment by using the piezocision. The secondary objectives are to evaluate the effect of this surgical technique on bone density, root resorption, osteoclast activity, inflammatory events and pain assessment. MATERIAL AND METHODS: The investigators will conduct a prospective study. The experimental group will consist of 14 adults, subjects from 18 to 40 years-old (10 women, 4 men). The control group will consist of 30 matched patients, who have been already treated in the orthodontic clinic of the University of Montreal. The reliabilities of Intra and Inter assesors will be measured for each doctor. After completion of the surgical guides from CBCT, the Piezocision will be performed the same day of the bracket indirect placement. The surgical procedure will be standardized and did it by the same surgeon. The appointments will be every 2 weeks for 4 months, then every month. The investigators will make an assessment of pain by using a numerical visual scale, during the first 7 days after surgery. Analysis of inflammatory markers (IL-1) and osteoclast activity (RANKL, OPG) will be evaluated from the gingival sulcus fluid collected at day 0, 1, 3, 5, 8, 12, 16 and 24 weeks. At the end of the treatment, the overall quality evaluation of treatment using the "American Board of Orthodontics' grading system" would be realized by two blind external observers to limit bias.

DETAILED DESCRIPTION:
EXPECTED RESULTS Orthodontic treatment accelerated by piézocicison will be completed within one year and will be 50% faster than a traditional treatment. The ratio benefit / risk of performing the piezocision will be acceptable for the patient and the orthodontist. We expect the following results: low pain, and absence of dental and periodontal deleterious effect (no root resorption, no tooth vitality loss and no bone loss). The same cohort can be used in future studies to assess the long term stability of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* normal or low skeletal problem;
* dental relationchip without extraction;
* healthy;
* complete adult teeth;
* very cooperative;
* no plaque;
* no active periodontal disease and no bone loss visible radiographically;
* patient wishing a shorter orthodontic treatment.

Exclusion Criteria:

* patient regularly taking analgesic and antidepressants.
* patients with alcool abuse problems.
* patient smoking more than 10 cigarettes per day.
* pregnant patient.
* allergy to non-steroidal anti-inflammatory drugs.
* local or systemic Immunodeficiencies.
* uncontrolled systemic disease (For exaemple diabetes, cardiovascular disease).
* coagulation problems or taking anti-coagulants.
* presence of oral infections and periodontal disease uncontrolled active.
* taking intravenous bisphosphonates or taking oral bisphosphonates for more than 4 years.
* taking a long-term corticosteroids.
* antibiotic necessary before any surgery and taking antibiotics within 6 months before surgery

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Determine the duration of orthodontic treatment associated with Piezocision | 18 months
  Assessment of the length of orthodontic treatment following piezocision

SECONDARY OUTCOMES:
Compare the duration of treatment with the control group | 18 months
  Compare the duration of treatment to the control group already processed and matched by sex, age, type of malocclusion, orthodontic biomechanics to limit bias.
Assess the overall quality of treatment (American Board of Orthodontics' grading system) | 18 months
  At the end of the treatment, the overall quality evaluation of treatment using the "American Board of Orthodontics' grading system" would be realized by two blind external observers to limit bias.
Assessment of pain during treatment (numerical visual scale) | Every days after the surgery durin 7 days and one day after every appointment
  Assessment of pain by Visual Digital Scale during treatment
Evaluation of osteoclastic activity (analysis of RANKL and OPG markers by sampling in the gingival fluid with sterile paper points) | weeks 0, 1, 3, 5, 8, 12, 16, 24
  Osteoclastic activity measurement by analysis of RANKL and OPG markers by sampling in the gingival fluid with sterile paper points
Evaluation of inflammatory markers (quantification of interleukin-1 (IL-1)) | weeks 0, 1, 3, 5, 8, 12, 16, 24
  Measurement of inflammatory markers in the gingival fluid with the quantification of interleukin-1 (IL-1)
Evaluate changes in density and bone volume with the cone beam computed tomography or Cone Beam Computerized Tomography (CBCT) | 18 months
  Evaluate changes in density and bone volume with the cone beam computed tomography or Cone Beam Computerized Tomography (CBCT)
Evaluate root resorption with the Cone Beam Computerized Tomography (CBCT) | 18 months
  Evaluation of root resorption using CBCT
Evaluate the inflammatory and remodelling gene expression | 0 and 8 weeks
  Evaluation of the gene expression associated with inflammation following piezocision

CONTACTS AND LOCATIONS:
Overall Officials: Julien Strippoli, DMD, Principal Investigator — University of Montreal, orthodontic department
Locations (1):
- University of Montreal, orthodontic department, Montreal, Quebec, Canada

REFERENCES:
- [Background] Brugnami F, Caiazzo A, Dibart S. Lingual orthodontics: accelerated realignment of the "social six" with piezocision. Compend Contin Educ Dent. 2013 Sep;34(8):608-10. PMID 24564613
- [Background] Dibart S, Sebaoun JD, Surmenian J. Piezocision: a minimally invasive, periodontally accelerated orthodontic tooth movement procedure. Compend Contin Educ Dent. 2009 Jul-Aug;30(6):342-4, 346, 348-50. PMID 19715011
- [Background] Dibart S, Surmenian J, Sebaoun JD, Montesani L. Rapid treatment of Class II malocclusion with piezocision: two case reports. Int J Periodontics Restorative Dent. 2010 Oct;30(5):487-93. PMID 20814602
- [Background] Dibart S, Yee C, Surmenian J, Sebaoun JD, Baloul S, Goguet-Surmenian E, Kantarci A. Tissue response during Piezocision-assisted tooth movement: a histological study in rats. Eur J Orthod. 2014 Aug;36(4):457-64. doi: 10.1093/ejo/cjt079. Epub 2013 Nov 19. PMID 24253033
- [Background] Keser EI, Dibart S. Piezocision-assisted Invisalign treatment. Compend Contin Educ Dent. 2011 Mar;32(2):46-8, 50-1. PMID 21473299
- [Background] Keser EI, Dibart S. Sequential piezocision: a novel approach to accelerated orthodontic treatment. Am J Orthod Dentofacial Orthop. 2013 Dec;144(6):879-89. doi: 10.1016/j.ajodo.2012.12.014. PMID 24286911
- [Background] Long H, Pyakurel U, Wang Y, Liao L, Zhou Y, Lai W. Interventions for accelerating orthodontic tooth movement: a systematic review. Angle Orthod. 2013 Jan;83(1):164-71. doi: 10.2319/031512-224.1. Epub 2012 Jun 21. PMID 22720793
- [Background] Milano F, Dibart S, Montesani L, Guerra L. Computer-guided surgery using the piezocision technique. Int J Periodontics Restorative Dent. 2014 Jul-Aug;34(4):523-9. doi: 10.11607/prd.1741. PMID 25006769
- [Background] Mathews DP, Kokich VG. Accelerating tooth movement: the case against corticotomy-induced orthodontics. Am J Orthod Dentofacial Orthop. 2013 Jul;144(1):5-13. doi: 10.1016/j.ajodo.2013.04.008. No abstract available. PMID 23810039
- [Background] Sebaoun JD, Surmenian J, Dibart S. [Accelerated orthodontic treatment with piezocision: a mini-invasive alternative to conventional corticotomies]. Orthod Fr. 2011 Dec;82(4):311-9. doi: 10.1051/orthodfr/2011142. Epub 2011 Nov 23. French. PMID 22105680
- [Background] Strippoli J, Aknin JJ. [Accelerated tooth movement by alveolar corticotomy or piezocision]. Orthod Fr. 2012 Jun;83(2):155-64. doi: 10.1051/orthodfr/2012015. Epub 2012 Jun 21. French. PMID 22717115
- [Background] Vercellotti T, Podesta A. Orthodontic microsurgery: a new surgically guided technique for dental movement. Int J Periodontics Restorative Dent. 2007 Aug;27(4):325-31. PMID 17726988
- [Background] Yamaguchi M. RANK/RANKL/OPG during orthodontic tooth movement. Orthod Craniofac Res. 2009 May;12(2):113-9. doi: 10.1111/j.1601-6343.2009.01444.x. PMID 19419454